CLINICAL TRIAL: NCT00702728
Title: A Study to Evaluate the Effectiveness of Induced Diuresis With Matched Hydration Therapy Compared to Standard Overnight Hydration in the Prevention of Contrast Induced Nephropathy -MYTHOS Study
Brief Title: Induced Diuresis With Matched Hydration Compared to Standard Hydration for Contrast Induced Nephropathy (CIN) Prevention
Acronym: MYTHOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Antonio Bartorelli, M.D., Centro Cardiologico Monzino- University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R100-CCFM S103/208; EUDRACT No: 2008-001200-23
Record Dates: First submitted 2008-06-11; First posted 2008-06-20 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2008-06

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast induced nephropathy; Furosemide; Percutaneous coronary interventions; Saline hydration
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Furosemide and matched saline hydration by RenalGuard system
  Interventions: Drug: Furosemide and matched saline hydration
- 2 (Active Comparator): Standard IV saline infusion
  Interventions: Drug: isotonic saline solution

INTERVENTIONS:
Drug: Furosemide and matched saline hydration — Subjects will begin treatment approximately 90 minutes prior to the start of catheterization procedure. After a pre-hydration bolus of 250 ml of normal saline solution over 30 minutes the patient will receive 0.5 mg/kg of furosemide intravenously. Then, a replacement solution (saline) is given in an amount matched (ml for ml) to the volume of urine produced. Matched hydration will occur prior, during, and 4 hours post procedure.
  Arms: 1
Drug: isotonic saline solution — Subjects will receive 1 ml/Kg/hr of intravenous saline solution for a minimum of 12 hours prior to catheterization. Hydration will continue to occur during the catheterization, and for a minimum of 12 hours post catheterization.
  Arms: 2

SUMMARY:
This study is being proposed with the objective to assess the potential benefits of induced diuresis by furosemide with matched hydration therapy compared to standard hydration in the prevention of contrast-induced nephropathy (CIN). It is expected that matched hydration will prove to be as effective as hydration alone, will avoid an overnight stay prior to the procedure, and thus will prove to be a less costly and more clinically manageable solution to the prevention of CIN.

DETAILED DESCRIPTION:
Radiocontrast agents (contrast) are widely used in coronary and peripheral vascular catheterization procedures. Although the use of these iodine-containing agents is vital for these procedures, it can be associated with adverse side effects. CIN is one of the most important adverse effects of contrast agents, and can cause substantial morbidity and mortality.

Although the exact mechanisms remain unknown, intravenous hydration before the catheterization procedure is the only current treatment that has been shown to reduce the incidence of CIN. However, in patients with baseline impairments in renal function, hydration is commonly performed at a rate significantly lower than that shown to provide protection due to the fear of overhydration and pulmonary edema. Previous studies have used diuretics to increase urine output and prevent overhydration. In addition to the benefit of increased urine flow, loop diuretics, such as furosemide, should be expected to provide additive benefit against another potential mechanism of CIN, medullary ischemia, as they reduce sodium reabsorption, and consequentially oxygen consumption, of the kidney. While the results of their use have been mixed, it appears that furosemide was deleterious in patients who became dehydrated, i.e. those in whom the urine output was substantially greater than the rate of hydration they received.

This problem may be overcome by a device, which is now available on the market, called the RenalGuard System. The System is capable of delivering saline solution to a patient in an amount matched to the volume of urine produced by the patient. The purpose of this matched fluid replacement is to prevent hypovolemia that may lead to hypotension or fluid overload.The aim of the study is to compare furosemide-induced diuresis with matched hydration therapy compared to standard hydration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female equal or greater than the age of 18 years old.
2. Scheduled to undergo a non-emergent catheterization procedure with anticipated to use ≥80 ml contrast media. Additional other procedure (e.g., left ventriculography, imaging of grafts, stenting, etc.) are allowable other than those listed below as exclusion criteria #1.
3. Subject is clinically stable for >24hrs defined as Killip Class 1
4. Baseline Renal Function eGFR < 60ml/min, by MDRD (Modification of Diet in Renal Disease) calculator.
5. Patient has agreed to all follow-up testing.

Exclusion Criteria:

1. Catheterization procedure requiring a direct renal injection of contrast or an injection into the descending aorta proximal to the renal arteries.
2. Requires emergent catheterization or primary percutaneous intervention.
3. Subject is anuric, has been hospitalized for any change in renal function or has undergone renal replacement therapy (hemodialysis or hemofiltration) within the past month.
4. Known inability to place a Foley catheter
5. Currently has a known electrolyte imbalance or clinically significant arrhythmias which compromise subject's hemodynamic state.
6. Has received intravenous contrast within 10 days of procedure or has a planned procedure using contrast within 72 hours following the procedure.
7. Has documented respiratory insufficiency as evidenced by an oxygen saturation of < 90% on room air assessed on day of procedure.
8. Currently receiving or expected to receive Mannitol or Lithium therapy
9. Planned addition, discontinuation or dose adjustment of the trimethoprim, cimetidine, metaclopramide and/or the use of non-steroidal anti-inflammatory drugs within 48 hours of the procedure.
10. Subject has a known hypersensitivity to furosemide.
11. Subject is currently, plans, or has been enrolled in another clinical study involving use of an investigational drug or device within the prior 30 days.
12. If female, subject is pregnant or breastfeeding.
13. Subject is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of CIN | 48-72 hours

SECONDARY OUTCOMES:
Blood chemistry, major adverse clinical events, safety | Hospitalizatiojn period

CONTACTS AND LOCATIONS:
Overall Officials: Antonio L Bartorelli, MD, Principal Investigator — University of Milan
Locations (1):
- Centro Cardiologico Monzino- University of Milan, Milan, Italy

REFERENCES:
- [Background] Marenzi G, Marana I, Lauri G, Assanelli E, Grazi M, Campodonico J, Trabattoni D, Fabbiocchi F, Montorsi P, Bartorelli AL. The prevention of radiocontrast-agent-induced nephropathy by hemofiltration. N Engl J Med. 2003 Oct 2;349(14):1333-40. doi: 10.1056/NEJMoa023204. PMID 14523141
- [Background] Mueller C, Buerkle G, Buettner HJ, Petersen J, Perruchoud AP, Eriksson U, Marsch S, Roskamm H. Prevention of contrast media-associated nephropathy: randomized comparison of 2 hydration regimens in 1620 patients undergoing coronary angioplasty. Arch Intern Med. 2002 Feb 11;162(3):329-36. doi: 10.1001/archinte.162.3.329. PMID 11822926
- [Background] Solomon R, Werner C, Mann D, D'Elia J, Silva P. Effects of saline, mannitol, and furosemide on acute decreases in renal function induced by radiocontrast agents. N Engl J Med. 1994 Nov 24;331(21):1416-20. doi: 10.1056/NEJM199411243312104. PMID 7969280
- [Background] Marenzi G, Lauri G, Campodonico J, Marana I, Assanelli E, De Metrio M, Grazi M, Veglia F, Fabbiocchi F, Montorsi P, Bartorelli AL. Comparison of two hemofiltration protocols for prevention of contrast-induced nephropathy in high-risk patients. Am J Med. 2006 Feb;119(2):155-62. doi: 10.1016/j.amjmed.2005.08.002. PMID 16443418
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Marenzi G, Ferrari C, Marana I, Assanelli E, De Metrio M, Teruzzi G, Veglia F, Fabbiocchi F, Montorsi P, Bartorelli AL. Prevention of contrast nephropathy by furosemide with matched hydration: the MYTHOS (Induced Diuresis With Matched Hydration Compared to Standard Hydration for Contrast Induced Nephropathy Prevention) trial. JACC Cardiovasc Interv. 2012 Jan;5(1):90-7. doi: 10.1016/j.jcin.2011.08.017. PMID 22230154